CLINICAL TRIAL: NCT03414515
Title: Endovascular Treatment of Peripheral Artery Disease.
Brief Title: Endovascular Treatment of Peripheral Artery Disease (PAD)
Status: Completed | Type: Observational
Sponsor: Duomed (Industry)
Responsible Party: Sponsor
Other Study IDs: BM-PAD--02
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Arterial Disease; Iliac Artery Disease; Femoropopliteal Occlusive Disease; Below-the-knee Obstruction
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with peripheral artery disease: located in the common and external iliac artery, the common and superficial femoral artery, the popliteal artery and/or the below-the-knee (BTK) arteries (anterior tibial artery, posterior tibial artery or peroneal artery).
  Interventions: Device: Endovascular intervention

INTERVENTIONS:
Device: Endovascular intervention — Endovascular treatment with stent or balloon according to current practice
  Other Names: Optimed Sinus Superflex 635; Qualimed Talor Minor; Cardionovum Legflow balloon 0.035 + 0.018 + 0.014; Optimed Nylotrack 0.035 + 0.018

SUMMARY:
The purpose of this observational study is to evaluate the performance and safety of endovascular treatment with stenting (Optimed Sinus Superflex 635 or Qualimed Pontos-pp) or balloon angioplasty (Cardionovum Legflow or Optimed Nylotrack .035 + .018) according to current practice. The goal of the study will be achieved by assessing binary restenosis with duplex ultrasound, peri- and postoperative complications, technical success, target lesion revascularization, amputation and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must sign the informed consent form prior to the index-procedure.
2. Patient is older than 18 years.
3. Patient is compliant with the requested follow-up visits at week 6 and month 12 and the treatment regime.
4. Patient suffers from mild to intermittent claudication (Rutherford 1-3) or critical limb ischemia (Rutherford 4-5).
5. Target lesion is an occlusion or diameter stenosis is ≥50% by visual estimate.
6. Target lesion is located in the common and external iliac artery, in the common and superficial femoral artery, popliteal artery and/or the below-the-knee (BTK) arteries (anterior tibial artery, posterior tibial artery or peroneal artery).

Exclusion Criteria:

1. Patients with Rutherford 0 and 6.
2. Patient is pregnant.
3. Patients with estimated Glomerular filtration rate (eGFR) < 30 mL/min/1.73m2.
4. Patient has an acute thrombus or aneurysm in the target arteries.
5. Patient has a life expectancy of <12 months.
6. Patient has a target lesion that cannot be crossed with a guidewire.
7. Patient suffers from acute limb ischemia defined as any sudden decrease in limb perfusion causing a potential threat to limb viability.
8. Patient has scheduled elective non-vascular procedures within 3 months after index-procedure. Vascular procedures are allowed within 3 months after the index-procedure if it is guaranteed that acetylic salicylic acid and clopidogrel intake is not interrupted.
9. Contraindication for anti-thrombotic therapy (coagulopathy, …).
10. Patient has a known intolerance to anti-thrombotic medication or contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral artery disease, located in the common and external iliac artery, the common and superficial femoral artery, the popliteal artery and/or the below-the-knee (BTK) arteries (anterior tibial artery, posterior tibial artery or peroneal artery).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Binary restenosis | at 12 months follow-up
  Binary restenosis defined as ≥ 50% re-obstruction of the target lesion will be assessed by duplex ultrasound (peak systolic ratio >2.4)

SECONDARY OUTCOMES:
Device-related complications | up to 12 months follow-up
  Registration of peri- and early/late postoperative complications
Immediate procedural outcome | during index-procedure
  The combination of technical success defined as a successful access and deployment of the device and achievement of a final residual diameter stenosis of <30% of the treated target lesion on the procedural completion angiography and procedural success defined as a combination of technical success and absence of procedural complications.
Clinical outcome | at baseline
  Rutherford classification
Clinical outcome | at 6 weeks follow-up
  Rutherford classification
Clinical outcome | at 12 months follow-up
  Rutherford classification
Primary sustained clinical improvement | at 12 months follow-up
  defined as sustained upward shift of ≥ 1 category on Rutherford classification without the need for repeated TLR in surviving patients.
Secondary sustained clinical improvement | at 12 months follow-up
  defined as sustained upward shift of ≥ 1 category on Rutherford classification including the need for repeated TLR in surviving patients.
Target lesion revascularization (TLR) | up to 12 months follow-up
  defined as an endovascular or surgical treatment due to a problem arising from the lesion (+1cm proximally and distally to include edge phenomena).
Mortality | up to 12 months follow-up
  Procedure-related and all-cause mortality.
Amputation | up to 12 months follow-up
  minor amputation defined as below the ankle and major defined as above the ankle.

CONTACTS AND LOCATIONS:
Locations (1):
- Heilig Hart Ziekenhuis, Mol, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No